CLINICAL TRIAL: NCT05118295
Title: Single Step Lesion Annotation and Localization of Suspicious Breast Lesions
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Administratively Complete
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2021-0842; NCI-2021-11361 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2021-10-13; First posted 2021-11-11 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Breast Lesions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- SAVI Scout® (Experimental): marker is accurately placed in the breast tumor
  Interventions: Device: SAVI Scout®

INTERVENTIONS:
Device: SAVI Scout® — Savi Scout marker is placed within 1 cm of the breast tumor

SUMMARY:
The SAVI Reflector is a nonradioactive infrared (IR)-activated electromagnetic wave device that can be implanted in the breast or lymph nodes under image-directed guidance, typically by mammography or sonography. Intraoperatively, the SCOUT hand-held device is then percutaneously applied to the breast or lymph node, creating an audible signal on the device console with a gradient which correlates to distance (in mm) from the target lesion and marker.

The Savi Scout surgical guidance system was approved by the U.S. Food and Drug Administration in 2014. Furthermore, it was approved for long term use, with no restrictions on the length of time in 2017.

The system consists of an implantable reflector with a 4-mm body size, preloaded in a 16-gauge deliverable needle, a hand-held probe and a console. The reflector consists of an IR light receptor, resistor switch and two antennae. This is placed into or near the target through a 16G needle under mammographic or sonographic guidance. The hand-held probe detects pulses of infrared (IR) light and radar wave signals, received by the console system, which then emits and receives signals back to the reflector to provide real time localization and target proximity information to the surgeon.

The SCOUT console provides audible and visual feedback intraoperatively, the frequency of which increases as the handheld reader approaches the implanted reflector. After excision of the breast lesion, the handheld reader can be used to immediately confirm removal of the reflector, present in the lumpectomy specimen, and subsequent quiescence of radar signal in the breast.

DETAILED DESCRIPTION:
Primary Endpoint:

-To measure success of surgical retrieval of SAVI Scout placed at the time of initial, or mid-chemo, imaging studies. To demonstrate the successful excision of unifocal tumor tissue and/or tumor bed (after neoadjuvant chemotherapy).

Other Endpoints:

* Safety: Number of device-related adverse events.
* Radiological Placement Radiologist-rated ease of placement using Likert scale
* Accuracy of placement:
* Accurate: Within the breast tumor
* Marginal: Within the peritumoral tissue < or equal 5 mm
* Inadequate: More than 5 mm
* Unacceptable: Required additional localization device placement
* Success rate of maintained position of SAVI Scout, measured on interval imaging:
* Accurate: Within the breast tumor
* Marginal: Within the peritumoral tissue < or equal 5 mm
* Inadequate: More than 5 mm

ELIGIBILITY:
Inclusion Criteria:

1. Female or male patients >18 years of age at the time of consent.
2. Unifocal BIRADS-5 or -6 lesions at the time of diagnostic imaging
3. Unifocal, histologically-proven T0-T3, N0-1 invasive breast cancer at the time of mid-chemotherapy imaging if receiving neoadjuvant therapy

Exclusion criteria

1. Distant metastasis
2. Inflammatory breast carcinoma
3. Nickel allergy
4. Patients with active cardiac implants
5. Patients participating in Protocol 2016-0046, Multicenter Trial for Eliminating Breast Cancer Surgery in Exceptional Responders to Neoadjuvant Therapy
6. Patients participating in Protocol AFT-25, Comparison of Operative to Monitoring and Endocrine Therapy for Low-risk DCIS (COMET)
7. Pregnant women will be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2022-04-11 (Actual); Primary Completion 2025-01-22 (Actual); Study Completion 2025-01-22 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v4.0, Change From Baseline in Pain Scores on the Visual Analog Scale at 6 Weeks | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Tanya Moseley, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: M D Anderson Cancer Center website — http://www.mdanderson.org